CLINICAL TRIAL: NCT05930067
Title: Continuation of Patient Follow-up to 2 Years for the Pinnacle RSA and Pinnacle DM RSA Clinical Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Radiostereometric Analysis Network (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS23122 - HS25079
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hip Osteoarthritis
Keywords: Hip Replacement
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Pinnacle Gription (Other): Pinnacle Gription Acetabular Cup
  Interventions: Device: Pinnacle Gription Acetabular Cup
- Pinnacle Dual Mobility (Other): Pinnacle Dual Mobility System
  Interventions: Device: Pinnacle Dual Mobility

INTERVENTIONS:
Device: Pinnacle Gription Acetabular Cup — Pinnacle Gription cup with Corail/ACTIS stem
  Arms: Pinnacle Gription
Device: Pinnacle Dual Mobility — Bi-Mentum AltrX liner
  Arms: Pinnacle Dual Mobility

SUMMARY:
The proposed study is a continuation of two prospective, multi-centre, non-controlled studies of the Pinnacle and Pinnacle Dual Mobility total hip arthroplasty systems, originally initiated by DePuy Synthes (DSJ_2018_02 and DJS_2019_02, respectively).

DETAILED DESCRIPTION:
The primary study objective is to establish the mean superior migration of the Pinnacle Gription Sector acetabular cup, irrespective of standard or dual mobility articulation, using model-based radiostereometric analysis. As both prior studies utilize the same acetabular component, a combined analysis will be performed with an additional sub-analysis on those with a Pinnacle Dual Mobility system. Additional objectives include comparison of acetabular cup migration between surgical approach groups (posterolateral, direct lateral, direct anterior) at all time points, linear head penetration at 1 and 2 years, as well as functional and health status outcomes. Patients will be followed to the original end point of 2 years post-surgery using the same radiographic and patient-reported outcome measures at the primary studies; Harris Hip Score, Hip Evaluation, HOOS Jr., and Forgotten Joint Score. Results of this study will be published in orthopaedic journals.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who were enrolled on the DSJ_2018_02 and DSJ_2019_02.

Exclusion Criteria:

1. Individuals have active local or systemic infection.
2. Individuals who have loss of musculature, neuromuscular compromise or vascular deficiency in the affected limb rendering the procedure unjustified.
3. Individuals with poor bone quality, such as osteoporosis, where in the surgeon's opinion, there could be considerable migration of the prosthesis or a significant chance of bone fracture and/or the lack of adequate bone to support the implant(s).
4. Individuals with Charcot's or Paget's disease.
5. Individuals who, in the judgement of the investigator, would not be a candidate for protocol allowable components to be used for their THA.
6. Women who are pregnant or lactating.
7. Individuals who have had a contralateral hip that was implanted less than 6 months prior to the time of consent into this study or individuals that expect to have a contralateral hip implanted in the 6 months following the time of consent into this study. Individuals that have amputations in either leg that would impact rehabilitation following surgery.
8. Individuals who are bedridden per the Investigators determination.
9. Individuals that have participated in a clinical investigation with an investigational product (drug or device) in the last three months.
10. Individuals currently involved in any personal injury litigation, medical-legal or worker's compensation claims.
11. Individuals, in the opinion of the Investigator, who are drug or alcohol abusers or have a psychological disorder that could affect their ability to complete patient reported questionnaires or be compliant with follow-up requirements.
12. Individuals diagnosed and taking prescription medications to treat a muscular disorder that limits mobility due to sever stiffness and pain such as fibromyalgia or polymyalgia.
13. Subject has a medical condition with less than 2 years life expectancy.
14. Individual has a BMI >45 kg/m2.
15. DSJ-2019-02 only: Individuals who require revision arthroplasty and have a well-fixed non-DePuy Synthes femoral stem or a well-fixed DePuy Synthes femoral stem that does not have a polished neck

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Changes in RSA Migrations from baseline(6-week) to 6-month, 1-year and 2-year | Post-op: 6-weeks, 3-months, 6-months, 1-year, 2-year
  Stability over a period of two year measured by migration (mm) with Röntgen Stereometric Analysis

SECONDARY OUTCOMES:
Subsidence profiles | 6-months, 1-year, 2-year
  Comparing RSA exams at the specified time points to determine relative movement of the device
Change of functional outcome over 2 year follow-up period (Harris Hip Score) | Preoperative, 6 weeks, 3 months, 6 months, 12 months and 2 years postoperatively
  The Harris Hip Score (HHS) is a score used in total hip arthroplasty, mainly combining range of motion questions with questions regarding daily life activities. The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. Results can be recorded and calculated online. The maximum score possible is 100, any result <70 is considered a poor result; The HHS is an outcome measure administered by a qualified health care professional.
Pain and Function | Preoperative, 6 weeks, 3 months, 6 months, 12 months and 2 years postoperatively
  The Hip Disability and Osteoarthritis Outcome score - joint replacement (HOOS JR) will be used. The HOOS-JR is a joint replacement survey designed to measure pain and function.
Forgotten Joint Score (FJS) | Preoperative, 6 weeks, 3 months, 6 months, 12 months and 2 years postoperatively
  The FJS total score range is 0-100, higher scores indicating the patient is able to forget the joint daily lower degree of joint awareness.
Complications | Preoperative, 6 weeks, 3 months, 6 months, 12 months and 2 years postoperatively
  Evaluate the type and frequency of the complications/adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Turgeon, MD, Principal Investigator — Concordia Joint Replacement Group
Locations (2):
- Canada (2):
  - Orthopaedic Innovation Centre, Winnipeg, Manitoba
  - London Health Sciences Centre, London, Ontario